CLINICAL TRIAL: NCT02170948
Title: The Analgesic Efficacy of Dexmedetomidine as a Local Anesthetic Adjunct in Ankle Blocks for Forefoot Surgery. A Dose Ranging Study.
Brief Title: The Effectiveness of the Addition of Dexmedetomidine to Analgesia for Ankle Surgery.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was very low
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-6795-A
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia
Keywords: ultrasound-guided regional anesthesia; nerve block; ankle block; dexmedetomidine; Precedex; ankle surgery; forefoot surgery; duration; anesthetic duration following ankle block for forefoot surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dex 0.5 (Experimental): Ropivacaine and Lidocaine plus Dexmedetomidine (0.5mg/kg) plus Normal Saline
  Interventions: Drug: Dexmedetomidine
- Dex 1.0 (Experimental): Ropivacaine and Lidocaine plus Dexmedetomidine (1.0mg/kg) plus Normal Saline
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — An anesthetic concoction of 2% Lidocaine, 1% Ropivacaine, and Dexmedetomidine diluted solution will be provided via a series of anesthetic injections related to the ankle block procedure
  Other Names: Precedex

SUMMARY:
Forefoot surgeries involve a relatively short operation usually completed in 1 - 1½ hours, with patients generally being allowed to go home on the same day. Despite this, post-surgery pain is often severe and a delay in the discharge of patients due to difficulty with pain control after the surgery is common.

Performing nerve blocks in association with sedation is the preferred way to provide pain relief and offers important benefits for foot surgeries. With nerve blocks, the requirement for oral painkillers and their associated side effects is reduced. Increasing the duration of local anesthetic action is helpful as it increases the time of pain relief, allowing for a smoother transition to oral pain medications, earlier discharge, and faster recovery.

Recently, Precedex has been considered for its usefulness in prolonging the pain relief produced by nerve blocks. The identified benefits of this particular use include reducing post-surgical pain medications requirements, reducing the incidence of nausea and vomiting, reducing the incidence of sedation from such medication, and diminishing the incidence of respiratory depression (inadequate breathing). Two small studies have also shown that adding dexmedetomidine to nerve block solution results in prolonging pain relief.

The purpose of the study is to examine several doses of dexmedetomidine combined with local anesthetic drugs and determine the best combination for prolonging pain relief, while minimizing potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* American Society of Anesthesiologists (ASA) I-III patients
* Ages 18-65
* Body Mass Index (BMI) ≤ 38 kg/m2

Exclusion Criteria:

* Preexisting neurological deficits or peripheral neuropathy in the distribution of the sciatic or femoral nerves
* Known coronary heart disease, congestive heart failure, cardiomyopathies, or arrhythmias
* Baseline line heart rate < 60 Beats Per Minute (BPM) or baseline systolic blood pressure < 100 mm Hg
* Medications that reduce heart rate
* Known liver or renal dysfunction or existing diseases affecting these organs
* Local infection
* Contraindication to regional anesthesia
* Chronic pain disorders
* History of use of over 30mg oxycodone or equivalent per day
* Contraindication to a component of multi-modal analgesia
* Allergy to local anesthetics or dexmedetomidine
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Inability to provide informed consent
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Duration of Analgesia | patients will be followed for two weeks
  Patients will be asked about the duration of their analgesia by asking when they first felt pain at the surgical site. Patients will be asked prior to discharge, and routinely during specified phone calls until analgesia wear off

SECONDARY OUTCOMES:
Requirements for pain medications; complications | weekly for up to 2 weeks
  Patients will be called at 24 hours, 7 days and 14 days and asked to describe their pain levels, the requirements for pain medication, and any complications that may have arisen post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada